CLINICAL TRIAL: NCT02979158
Title: Influence of Cardiopulmonary Bypass on Platelet Function in Patients With Preoperative Dual Antiplatelet Therapy:
Brief Title: Preoperative Dual Antiplatelet Therapy: Platelet Function and Influence of Cardiopulmonary Bypass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DAPTUMU-123
Record Dates: First submitted 2016-11-21; First posted 2016-12-01 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2016-11

CONDITIONS: Cardiopulmonary Bypass; Platelet Disorder; Bleeding Disorder; Platelet Dysfunction Due to Drugs
MeSH Terms: conditions — Blood Platelet Disorders; Hemostatic Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CPB Low Dose (Experimental): Conduct of cardiopulmonary bypass using a low heparin dose verified by the activated clotting time at 250 s
  Interventions: Procedure: CPB Low Dose
- CPB High Dose (Experimental): Conduct of cardiopulmonary bypass using a high heparin dose verified by the activated clotting time at 480 s
  Interventions: Procedure: CPB High Dose

INTERVENTIONS:
Procedure: CPB Low Dose — Performing CPB with low dose heparin and coated equipment
  Arms: CPB Low Dose
Procedure: CPB High Dose — Performing CPB with high dose heparin and uncoated equipment
  Arms: CPB High Dose

SUMMARY:
Patients admitted for coronary artery bypass surgery taking antiplatelet medicine have an increased risk for bleeding.

Present study aims to compare the platelet function in two patient groups using different types of heart-lung machine methods.

It is assumed that one of the methods is superior verified by sensitive methods of testing platelet function.

DETAILED DESCRIPTION:
Taking antiplatelet medication before cardiac surgery increases the risk for bleeding.

The surgical procedure and the use of a heart-lung machine may disturb the function of platelets, why measures to protect the existing function of platelets are of prime concern.

The present study aims to compare how two types of heart-lung machine methods influence platelet function in two groups of patients.

The platelet function will be tested before, during and after surgery by the use of two independent methods.

ELIGIBILITY:
Inclusion Criteria:

* Patients accepted for coronary bypass surgery with dual preoperative antiplatelet therapy suspended less than 4 days prior to surgery

Exclusion Criteria:

* Abnormal coagulation verified from preoperative assessments, platelet count <100 000, Warfarin medication and renal insufficiency (GFR < 60 ml/min)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-11; Primary Completion 2018-01-24 (Actual); Study Completion 2018-01-24 (Actual)

PRIMARY OUTCOMES:
Assessment of platelet function following cardiopulmonary bypass using platelet aggregometry | Test of platelet function will be analysed on arrival to the operating room, post cardiopulmonary bypass and on day 1 in the intensive care unit based on the area under the curve depited from the two employed aggremometers
  Included aggregometry tests: Multiplate and Rotem Platelet

SECONDARY OUTCOMES:
Postoperative bleeding | Postoperative bleeding 24 hrs
  Blood loss 24 hrs post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Näslund, MD PhD, Principal Investigator — Department of Publich Health and Clinical Medicin, Umeå University, Sweden; Magnus Hedström, MD, Study Director — Heart Centre Umeå University Hospital Sweden
Locations (1):
- Heart Centre Umeå University Hospital, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared after reviewing final results after study completion at this site and through publication in a scientific journal.

REFERENCES:
- [Background] Olsson A, Alfredsson J, Hakansson E, Svedjeholm R, Berglund J, Berg S. Protamine reduces whole blood platelet aggregation after cardiopulmonary bypass. Scand Cardiovasc J. 2016;50(1):58-63. doi: 10.3109/14017431.2015.1099720. Epub 2015 Oct 20. PMID 26402229
- [Background] Mishra PK, Thekkudan J, Sahajanandan R, Gravenor M, Lakshmanan S, Fayaz KM, Luckraz H. The role of point-of-care assessment of platelet function in predicting postoperative bleeding and transfusion requirements after coronary artery bypass grafting. Ann Card Anaesth. 2015 Jan-Mar;18(1):45-51. doi: 10.4103/0971-9784.148321. PMID 25566711
- [Background] Mollnes TE, Videm V, Christiansen D, Bergseth G, Riesenfeld J, Hovig T. Platelet compatibility of an artificial surface modified with functionally active heparin. Thromb Haemost. 1999 Sep;82(3):1132-6. PMID 10494777